CLINICAL TRIAL: NCT00903305
Title: A Standard Nursing Intervention Protocol for Breast Cancer as a Chronic Illness
Brief Title: Nurse-Provided Care or Standard Care in Treating Patients With Stage I, Stage II, or Stage III Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR0000629408; P30CA033572 (NIH); CHNMC-08031
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Fatigue; Nausea and Vomiting; Pain
Keywords: pain; fatigue; nausea and vomiting; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Nausea; Vomiting; Pain | interventions — Therapeutics; Psychiatric Rehabilitation

ARMS (2):
- Group II (SNIP) (Experimental): Patients undergo SNIP comprising four visits over 2 months and four monthly telephone calls from the APN. The APN will provide 24 hour access during the study. Patients complete questionnaires about satisfaction with care, perceived preparedness with self-care, and helpfulness of patient teaching at baseline, 3 months and 6 months.
  Interventions: Other: medical chart review; Other: questionnaire administration; Procedure: fatigue assessment and management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment
- Group I (usual care intervention) (Active Comparator): Patients undergo usual care and complete questionnaires about satisfaction with care, perceived preparedness with self-care, and helpfulness of patient teaching at baseline, 3 months and 6 months.
  Interventions: Other: medical chart review; Other: questionnaire administration; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: fatigue assessment and management
Procedure: psychosocial assessment and care
  Arms: Group II (SNIP)
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Meeting with a nurse to assess symptoms and quality of life may be more effective than standard care in treating patients with breast cancer.

PURPOSE: This clinical trial is studying nurse-provided care to see how well it works compared with standard care in treating patients with stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the effects of an advanced practice nurse, standardized nursing intervention protocol (SNIP) model vs usual care on overall quality of life and psychological distress of patients with stage I-III breast cancer, from initial treatment to 6 months post diagnosis.
* To compare symptom control in these two groups.
* To compare geriatric assessment outcomes in these two groups.
* To test the effects of the SNIP intervention as compared to the usual care group on resource use by these patients.
* To test the effects of SNIP on patients' and clinicians' satisfaction with care.
* To describe the effects of SNIP on patients' management of transitions from one phase of chronic illness to another.
* To identify subgroups of these patients who benefit most from the SNIP in relation to sociodemographic characteristics, disease/treatment factors, and geriatric assessment predictors.
* To obtain feedback from clinicians regarding interpretation of findings and application to the routine care of breast cancer patients.

OUTLINE: Patients are enrolled sequentially to 1 of 2 groups. Group 1 is enrolled during months 4-21 and group 2 is enrolled during months 25-54.

* Group 1 (usual care): Patient questionnaires are administered at baseline and at 3 and 6 months. The clinicians' satisfaction with care is also evaluated.
* Group 2 (advanced practice nurse [APN] intervention): Patients are accrued by an APN. Patients meet with the APN periodically to assess their physical well-being including ambulatory care needed, care of physical symptoms (i.e., pain, fatigue, nausea and vomiting), and psychological well-being. Questionnaires are administered at baseline and at 3 and 6 months.

In both groups, questionnaires include the FACT-Breast, Memorial Symptom Assessment Scale, Psychological Distress Thermometer, Comprehensive Geriatric Assessment, and Patient Satisfaction with Intervention. Clinicians also complete questionnaires. Patients' medical charts are also reviewed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I, II, or III breast cancer
* Admitted to City of Hope National Medical Center

  * Resides within a 30-mile radius of the medical center
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No prior cancer

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Quality of life, psychological distress, symptom relief, geriatric assessment outcome, and resource use at 3 months
Long-term impact at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSc, FAAN, Principal Investigator — City of Hope Comprehensive Cancer Center